CLINICAL TRIAL: NCT02946333
Title: Observational Study to Assess Disease Burden, in Terms of Health-related Quality of Life and Direct Healthcare Costs, in Patients With Newly Diagnosed Multiple Myeloma Who Are Not Candidates for Autologous Stem Cell Transplant (ASCT) in Spain
Brief Title: A Study to Assess Disease Burden, in Terms of Health-related Quality of Life and Direct Healthcare Costs, in Patients With Newly Diagnosed Multiple Myeloma Who Are Not Candidates for Autologous Stem Cell Transplant (ASCT) in Spain
Acronym: QoLMMBuS
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CEL-MIE-2016-01
Record Dates: First submitted 2016-09-30; First posted 2016-10-27 (Estimated); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; autologous stem cell transplant (ASCT); QoLMMBuS; healthcare costs
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient with MM who are not candidates for ASCT: Patients with newly diagnosed MM who are not candidates for ASCT and who are going to start drug treatment for the study disease and patient who is capable of understanding and filling in the study questionnaires At least 450 patients will be enrolled in a 2-year period. Patients must meet all of the inclusion criteria and none of the exclusion criteria and must have previously granted their informed consent in writing.

SUMMARY:
Those patients with newly diagnosed Multiple Myeloma (MM) who are not candidates for Autologous Stem Cell Transplant (ASCT) and who meet the screening criteria described in this protocol can participate. The participating patients must sign an informed consent, which the investigator who will collect the study variables in an electronic case report form (eCRF) will provide to them. The investigators must recruit at least 450 patients in a 24-month period.

DETAILED DESCRIPTION:
Following the baseline enrolment visit, the following data corresponding to the patient's visits scheduled according to routine clinical practice will be collected in accordance with the following model:

1. Recruitment period: data collection at the baseline visit, every 4 months +/- 15 days in the first year (month 4, 8 and 12) and every 6 months +/- 1 month in the second year (month 18 and 24).
2. Follow-up period: (study will end at 4 years following enrolment of the first patient)

   * From month 24 until up to 4 years from enrolment of the first patient, follow-ups will be performed with semi-annual data collections coinciding with the patient's routine clinical practice visits.
   * In case of progression, suspension or unexpected termination of treatment (for example due to toxicity), or death, a data collection coinciding with the visit in which any of the cases presented occurs will be performed.
   * If a new line of treatment is started, the follow-up model will be started with the same frequency of follow-ups described in point 1 above (month 4, 8, 12, 18 and 24 and semi-annually according to routine clinical practice until up to 4 years from enrolment of the first patient in the study).
3. Observation period: Following this 4-year period, an additional 5-year follow-up will be performed only to evaluate the onset of second primary malignant neoplasms. This follow-up during the 5-year observational period will be performed semi-annually (± 1 month) according to routine clinical practice at each site.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age.
* Patient with newly diagnosed multiple myeloma (MM) according to IMWG criteria who are not candidates for ASCT and who start treatment for the study disease.
* Patient who is capable of understanding and filling in the study questionnaires.
* Patient who has granted his or her informed consent in writing.

Exclusion Criteria:

* Patient who is participating in the active phase of treatment of any clinical trial during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 450 patients with newly diagnosed multiple myeloma (MM) according to IMWG criteria who are not candidates for ASCT and who start drug treatment for the study disease will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2016-12-25 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life (HRQoL) | 4 years
  This questionnaire consists of 30 items grouped into 8 dimensions: number of drugs, gait velocity, mood, activities of daily living, health status, nutrition, mental state and comorbidity/habits. It is an instrument that was developed and validated to assess the health status of elderly patients diagnosed with different hematological diseases, including MM. This scale may be a useful instrument in clinical practice as a support tool to predict tolerance to treatment in advanced age. The time required to complete the questionnaire is approximately 10-12 minutes. It will be provided only at the baseline visit for the patient to fill in before starting treatment. The patient must fill it in again each time he or she starts a new line. The questionnaire will be provided by the physician during the visit.
EuroQoL 5-Dimension, 5-Level Questionnaire (EQ-5D-5L) | 4 years
  This is a generic HRQoL questionnaire that contains a descriptive system and a visual analogue scale (VAS) for self-assessment of health status. The EQ-5D-5L's descriptive system contains a description of health state in five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has 5 possible responses. The respondent must mark the level of problems, within each dimension, that best describes his or her health state "today". It will be provided at each visit for the patient to fill in before starting treatment: at the baseline visit, approximately every 4 months in the first year (the visits must coincide with the patient's routine clinical practice visit) and after the first year every 6 months to progression. In case of progression and start of a second line of treatment, the questionnaire will start to be filled in with the same frequency initially described (baseline, every 4 months, etc.).
Quality of Life Questionnaire (QLQ-C30) | 4 years
  This is a cancer-specific questionnaire that consists of 30 items structured into 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning and social functioning), 3 symptom scales (fatigue, nausea and vomiting, pain), a global health status scale and, finally, 6 independent items (dyspnoea, insomnia, appetite loss, constipation, diarrhea and financial difficulties). Values from 1 to 4 are assigned depending on the patient's responses to the item. Only items 29 and 30 are evaluated with scoring from 1 to 7. Scores are standardised to obtain a score from 0 to 100, which determines the level of impact of the cancer on the patient for each scale. High scores on the overall health and functional status scales indicate a better QoL, while high scores on the symptoms scale would indicate a decrease in QoL since they indicate the presence of cancer-related symptoms.
Quality of Life Questionnaire - Multiple Myeloma Module 20 (QLQ-MY20) | 4 years
  This is a specific questionnaire used in combination with the QLQ-C30 generic questionnaire to evaluate quality of life in patients with MM. It consists of 20 items that address four specific domains - disease symptoms, side effects of treatment, future perspective and body image - and analyses various aspects of each dimension. Three of the four domains of the QLQ-MY20 are multi-item scales: Disease symptoms , side effects of treatment and future perspective (includes worry about death and health in the future and thinking about illness). The body image scale is a single-item scale that addresses physical attractiveness. The scores obtained are transformed linearly to a scale from 0 to 100. A high score in the disease symptoms and side effects domains represents a high level of symptoms or problems, while a high score in the future perspective and body image domains represents better outcomes.
Health care cost for Multiple Myeloma (MM) patients | 4 years
  MM-related direct healthcare resources and costs will be evaluated in each line MM treatment will be evaluated. The questionnaire will be provided by the physician during the visit. The resources used since the previous study visit will be collected at each visit.

SECONDARY OUTCOMES:
Time to progression (TTP) | 4 years
  Time that elapses from the start of a treatment up to disease progression.
Progression-free survival (PFS) | 4 years
  Time that elapses from the start of a treatment to disease progression or death, whichever occurs first.
Overall survival (OS) | 9 years
  Time that elapses from the diagnosis of the disease up to the death of the patient for any reason.
Overall response rate | 4 years
  Response measured through the IMWG criteria: Stringent complete response; complete response (CR); very good partial response; partial response (PR); stable disease (SD); progression (P)
Response duration | 4 years
  For each line of treatment for multiple myeloma (MM) during the study period
Treatment-free interval [TFI] | 4 years
  Time between relapse and start of a new treatment (second/third lines)

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Lostaunau, Senior Medical Advisor MM, Study Director — Celgene
Locations (65):
- Spain (65):
  - Hospital Punta de Europa, Algeciras, Andalusia
  - Hospital de Antequera, Antequera, Andalusia
  - Hospital Reina Sofía, Córdoba, Andalusia
  - Hospital Huercal Olvera, Huercal Olvera, Andalusia
  - Hospital General Jaén, Jaén, Andalusia
  - Hospital Jerez de la Frontera, Jerez de la Frontera, Andalusia
  - Clinico Univ. Virgen de la Victoria, Málaga, Andalusia
  - Hospital Carlos Haya, Málaga, Andalusia
  - Hospital de Costa del Sol, Málaga, Andalusia
  - Hospital de Motril, Motril, Andalusia
  - Hospital Valle de los Pedroches Pozoblanco, Pozoblanco, Andalusia
  - Hospital Puerto Real, Puerto Real, Andalusia
  - Hospital de Macarena, Seville, Andalusia
  - Hospital Miguel Servet, Zaragoza, Aragon
  - Hospital Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Hospital ICO Durán y Reynals, L'Hospitalet de Llobregat, Barcelona
  - ICO Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Basurto, Bilbao, Basque Country
  - Hospital de Galadakao, Usansolo, Basque Country
  - Hospital de Txagorritxu, Vitoria-Gasteiz, Basque Country
  - Hospital Universitario Dr. Negrín, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Dr. Negrín, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife, Canary Islands
  - Hospital Universitario de Burgos, Burgos, Castille and León
  - Hospital Clínico Universitario de Salamanca, Salamanca, Castille and León
  - Hospital Clínico de Valladolid, Valladolid, Castille and León
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Vall Hebrón, Barcelona, Catalonia
  - Hospital General de Granollers, Granollers, Catalonia
  - Hospital Arnau Vilanova de Lleida, Lleida, Catalonia
  - Fundació Althaia, Manresa, Catalonia
  - Parc Taulí, Sabadell, Catalonia
  - Mutua Terrassa, Terrassa, Catalonia
  - Complejo Hospitalario Llerena-Zafra, Llerena, Extremadura
  - Hospital de Mérida, Mérida, Extremadura
  - Complexo Hospitalario Universitario de A Coruña, A Coruña, Galicia
  - Hospital Lucus Augustí, Lugo, Galicia
  - Complexo Hospitalario Universitario de Ourense, Ourense, Galicia
  - Complexo Hospitalario de Pontevedra, Pontevedra, Galicia
  - Complexo Hospitalario Universitario de Vigo, Vigo, Galicia
  - Hospital Universitario Canarias, Santa Cruz de Tenerife, Islas Canaria
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital de la Princesa, Madrid, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Quirón, Pozuelo de Alarcón, Madrid
  - Hospital Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Complejo Hospitalario de Navarra, Navarra, Navarre
  - Complejo Hospitalario Navarra, Pamplona, Navarre
  - Hospital de La Ribera, Alzira, Valencia
  - Hospital General Castellón, Castellon, Valencia
  - Hospital Arnau Vilanova Valencia, Valencia, Valencia
  - Hospital Doctor Peset, Valencia, Valencia
  - Hospital La Fe Valencia, Valencia, Valencia
  - Hospital La Ribera, Valencia, Valencia
  - Complejo Hospitalario de Ávila, Ávila
  - Hospital Infanta Leonor, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital La Paz, Madrid
  - Hospital Universitario La Fe, Valencia
  - Hospital Miguel Servet, Zaragoza

REFERENCES:
- [Derived] Engelhardt M, Ihorst G, Singh M, Rieth A, Saba G, Pellan M, Lebioda A. Real-World Evaluation of Health-Related Quality of Life in Patients With Multiple Myeloma From Germany. Clin Lymphoma Myeloma Leuk. 2021 Feb;21(2):e160-e175. doi: 10.1016/j.clml.2020.10.002. Epub 2020 Oct 24. PMID 33218965